CLINICAL TRIAL: NCT05010356
Title: Study of Molecular Causes of Metabolic Disorders in Obese Premenopausal Women After Breast Cancer
Brief Title: Insulin Sensitivity After Breast Cancer
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Copenhagen (Other)
Responsible Party: Principal Investigator, Lykke Sylow, Associate Professor, University of Copenhagen
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 514-0213/21-5000
Record Dates: First submitted 2021-06-23; First posted 2021-08-18 (Actual); Last update posted 2021-08-18 (Actual); Status verified 2021-08

CONDITIONS: Insulin Sensitivity/Resistance; Breast Cancer; Survivorship; Metabolic Disturbance
MeSH Terms: conditions — Insulin Resistance; Breast Neoplasms | interventions — Insulin

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Healthy control subjects (Experimental): Healthy control subjects undergoing a hyperinsulinemic euglycemic clamp
  Interventions: Drug: Insulin
- Breast cancer survivors (Experimental): Breast cancer survivors undergoing a hyperinsulinemic euglycemic clamp
  Interventions: Drug: Insulin

INTERVENTIONS:
Drug: Insulin — Hyperinsulinemic euglycemic clamp
  Other Names: Hyperinsulinemic euglycemic clamp

SUMMARY:
Epidemiological studies have revealed that 60-80% of women with breast cancer (BC) develop metabolic disorders that are similar to those observed in conditions like type 2 diabetes. These metabolic disorders, including insulin resistance, obesity, hyperinsulinemia, and glucose intolerance, are associated with increased BC recurrence and mortality. Skeletal muscle is the major site of glucose uptake in humans. The aims of the present project are to 1) determine the involvement of insulin resistance in skeletal muscle in the metabolic disorders prevalent in BC survivors, 2) identify BC-and/or treatment-induced molecular changes in skeletal muscle from BC survivors .

DETAILED DESCRIPTION:
Up to 80% of women with breast cancer (BC) develop metabolic disorders, such as insulin resistance, obesity, hyperinsulinemia, and glucose intolerance, during or after their treatment. Such disorders increase BC mortality and the likelihood of relapse 2- and 3-fold, respectively. However, it is not known why BC and/or the treatment hereof causes metabolic disorders and very few studies have investigated the underlying biological causes.

Aims:

1. determine the involvement of insulin resistance in skeletal muscle in the metabolic disorders prevalent in BC survivors
2. identify BC-and/or treatment-induced molecular changes in skeletal muscle

BC is a common cancer with 2.1 million new cases each year, and BC also causes the largest number of cancer-related deaths among women worldwide. Fortunately, more people are now surviving their cancer. In Denmark, the majority of the 300.000 cancer survivors, constitute a group of ~ 70,000 women who have survived BC. However, there is a severe lack of research into the physiological sequelae of cancer and/or treatment, including the metabolic health consequences of BC. Recent epidemiological studies have revealed that 60-80% of women with BC develop metabolic disorders that are similar to those observed in conditions such as type 2 diabetes (T2D) during or following their treatment. However, unlike T2D, the underlying biological causes for the development of metabolic disorders with BC and/or the treatment are poorly investigated. It is important to address this knowledge gap, as metabolic disorders increase mortality among women with BC 2-fold and increase the likelihood of BC recurrence up to 3-fold.

The investigators hypothesize that metabolic disorders in BC survivors are due to cancer and/or treatment-mediated molecular rewiring of skeletal muscle, which causes insulin resistance.

Scientific breakthroughs in obesity and diabetes research have shown that hyperinsulinemia and hyperglycemia are most often caused by insulin resistance in skeletal muscle, fat, and liver. In particular, skeletal muscle is essential for maintaining a normal metabolism as it is responsible for up to 75% of the uptake of glucose from the blood in response to insulin. It is thus likely that skeletal muscle insulin resistance causes metabolic perturbations in BC survivors but this has not been investigated directly. Insulin-resistant skeletal muscle does not respond normally to insulin, causing severe metabolic disorders. These include hyperglycemia, hyperinsulinemia, dyslipidemia and hypertension; all conditions that are increasingly being documented in women with BC and BC survivors It is likely that insulin resistance in skeletal muscle is causing the metabolic disorders often present in BC survivors. Since muscle plays key roles in metabolic regulation by keeping blood glucose and insulin levels normal, it is extremely relevant to clarify the precise involvement of skeletal muscle in BC-related metabolic disorders.

12 premenopausal women (Body Mass Index = 25-30) who were operated for BC (stage I-III) will be included. Especially overweight premenopausal women develop markedly metabolic dysfunction as determined by an oral glucose tolerance test. The subjects will be studied 3-10 weeks after completing adjuvant chemotherapy. Twelve healthy weight-, activity- and age-matched subjects will be recruited as controls (matched by bicycle exercise test, grip strength, dual x-ray absorptiometry, and using the international physical activity questionnaire). Exclusion criteria are as follows: Post-menopause at the time of BC diagnosis, metastatic cancer, < 4 or > 5 series of paclitaxel treatment, alcohol intake of > 7 items/week, smoking, known T2D or metabolic syndrome, known cardiovascular disease and medical treatment thereof, or impaired mobility. Insulin sensitivity will be measured via the hyperinsulinemic-euglycemic clamp method. In short, basal muscle (from the vastus lateralus muscle) biopsies are taken after 1 hour rest after which insulin (1.4 mU/kg/min) is administered while maintaining euglycemia by continuous glucose infusion. Insulin-stimulated biopsies are taken after 1.5 hours.

ELIGIBILITY:
Inclusion Criteria:

* Premenopausal women operated for breast cancer and after completing adjuvant chemotherapy and no earlier than 3 weeks after its termination
* BMI: 25-30
* Healthy controls will be included matched by gender, weight, age, and level of physical activity to the patient group included as subjects

Exclusion Criteria:

* Known postmenopause occurred at the time of diagnosis of breast cancer
* Alcohol intake of> 7 items / week
* Smoker
* Already known Type 2 diabetes mellitus or metabolic syndrome and medical treatment thereof.
* Cardiovascular disease and its medical treatment
* Impaired mobility

Ages: 20 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Estimated)
Dates: Start 2021-08 (Estimated); Primary Completion 2022-12 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Insulin sensitivity status | 2 years
  Glucose infusion rate during the hyperinsulinemic euglycemic clamp to ascertain the insulin sensitivity
Hepatic glucose production | 2 years
  Measurements from the Hyperinsulinemic Euglycemic Clamp will be used to assess insulin effects on hepatic glucose production

SECONDARY OUTCOMES:
Proteomic changes in skeletal muscle | 4 years
  Skeletal muscle biopsies from the vastus lateralis muscle will be analysez using mass spectometry to determine proteomic chances in response to breast cancer in skeletal muscle
Insulin signaling | 4 years
  Intracellular insulin signaling will be determined using western blotting technique

CONTACTS AND LOCATIONS:
Overall Officials: Lykke Sylow, PhD, Principal Investigator — University of Copenhagen
Locations (1):
- University of Copenhagen, Copenhagen, DK, Denmark

IPD SHARING:
Plan to Share IPD: No